CLINICAL TRIAL: NCT01879579
Title: The Mobile Insulin Titration Intervention (MITI) Study: Innovative Chronic Disease Management of Diabetes
Brief Title: Mobile Insulin Titration Intervention
Acronym: MITI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Natalie Levy, Assistant Professor of Medicine, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S12-03713; UL1TR000038 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus
Keywords: Insulin; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile Insulin Titration Intervention (Experimental): Mobile Insulin Titration Intervention (MITI) arm patients will relay their fasting blood glucose levels to the study staff via text message. The patient will receive insulin titration instructions through a weekly phone call with a diabetes nurse.
  Interventions: Other: Mobile Insulin Titration Intervention
- Current Best Practice (No Intervention): Current Best Practice (CBP) arm patients will be treated according to the current best practice of insulin titration. They will attend scheduled clinic visits during which the provider will review their blood glucose logs and provide insulin titration instructions.

INTERVENTIONS:
Other: Mobile Insulin Titration Intervention — Patients send their fasting blood glucose levels to the clinic diabetes nurses via text message each weekday. The diabetes nurses call each patient once a week to give insulin titration instructions to replace in-person clinic visits for insulin titration.
  Arms: Mobile Insulin Titration Intervention

SUMMARY:
The purpose of this pilot study is to determine whether text message (and phone) communication can be effectively utilized to adjust long-acting insulin, compared to standard practice.

DETAILED DESCRIPTION:
The current practice of insulin titration for diabetics requires multiple in-person clinic visits, during which a patient's long-acting insulin dose is adjusted until the optimal dose to control glycemia is reached. Finding this optimal dose can take weeks in an ideal setting, but often takes much longer in a busy urban clinic such as Bellevue Hospital Center. Relaying titration instructions to patients via phone and text message has the potential to decrease the titration timeline, thus reducing the number of clinic visits and the time it takes patients to reach their target blood glucose levels.

For this pilot project, study staff will recruit patients who are initiating long-acting insulin treatment or initiating the titration of their existing long acting insulin treatment at Bellevue Hospital Center's Adult Primary Care Center. Patients who volunteer to enroll and provide informed consent will be randomized to one of two arms (MITI or current best practice arm) at the time of enrollment and stratified by whether the patient is initiating insulin treatment or initiating the titration of his/her existing insulin dose. The study staff will provide a cell phone (for temporary use) to any patients who are randomized to the MITI arm and don't own a personal cell phone (or whose personal cell phone is not able to receive the Sense Health text messages). Patients will use the cell phone free of cost to participate in the intervention (receive Sense Health text messages, send their fasting blood glucose levels, and speak with the diabetes nurse and study staff.)

Patients in the MITI arm will receive automated text messages 5 weekdays per week, for up to 12 weeks, from Sense Health. These text messages will request the patient's fasting blood glucose level. The patient will reply with his/her fasting blood glucose value, which will be logged in password-protected accounts on www.sensehealth.com. The clinic's diabetes nurses will check each patient's fasting blood glucose level on www.sensehealth.com each weekday and call any patient with fasting blood glucose values < 80 mg/dL and > 400 mg/dL. Each Thursday, patients will receive a phone call from a nurse, who will adjust the patient's insulin dose according to the study titration protocol. Each patient will continue to receive daily text messages and weekly phone calls until the first of three events occur: the patient reaches his/her optimal insulin dose for achieving glycemic control, 12 weeks elapse, or the patient withdraws from the study.

Patients in the current best practice arm (CBP) will attend scheduled clinic appointments during which a provider will review the patient's fasting blood glucose log and titrate the insulin dose according to current best practice.

Patients in both arms will continue receiving routine care, including HbA1c values every 3 months and other routine labs and measures as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Initiating long-acting insulin treatment or initiating the titration of long-acting insulin treatment
* Speaks English or Spanish
* Hemoglobin A1c > or = 8%
* Able and willing to inject insulin
* Able and willing to provide informed consent

Exclusion Criteria:

* Short-acting insulin treatment
* Systemic glucocorticoids
* Sustained elevated serum creatinine > or = 1.5 mg/dL for men and > or = 1.4 mg/dL for women
* Hypoglycemia unawareness
* Type 1 diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Levy, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Adult Primary Care Clinic, Bellevue Hospital Center, New York, New York, United States

REFERENCES:
- [Background] Riddle MC, Rosenstock J, Gerich J; Insulin Glargine 4002 Study Investigators. The treat-to-target trial: randomized addition of glargine or human NPH insulin to oral therapy of type 2 diabetic patients. Diabetes Care. 2003 Nov;26(11):3080-6. doi: 10.2337/diacare.26.11.3080. PMID 14578243
- [Background] Davies M, Storms F, Shutler S, Bianchi-Biscay M, Gomis R; ATLANTUS Study Group. Improvement of glycemic control in subjects with poorly controlled type 2 diabetes: comparison of two treatment algorithms using insulin glargine. Diabetes Care. 2005 Jun;28(6):1282-8. doi: 10.2337/diacare.28.6.1282. PMID 15920040
- [Background] Davies M, Lavalle-Gonzalez F, Storms F, Gomis R; AT.LANTUS Study Group. Initiation of insulin glargine therapy in type 2 diabetes subjects suboptimally controlled on oral antidiabetic agents: results from the AT.LANTUS trial. Diabetes Obes Metab. 2008 May;10(5):387-99. doi: 10.1111/j.1463-1326.2008.00873.x. Epub 2008 Mar 18. PMID 18355327
- [Background] Blonde L, Merilainen M, Karwe V, Raskin P; TITRATE Study Group. Patient-directed titration for achieving glycaemic goals using a once-daily basal insulin analogue: an assessment of two different fasting plasma glucose targets - the TITRATE study. Diabetes Obes Metab. 2009 Jun;11(6):623-31. doi: 10.1111/j.1463-1326.2009.01060.x. PMID 19515182
- [Background] Arora S, Peters AL, Agy C, Menchine M. A mobile health intervention for inner city patients with poorly controlled diabetes: proof-of-concept of the TExT-MED program. Diabetes Technol Ther. 2012 Jun;14(6):492-6. doi: 10.1089/dia.2011.0252. Epub 2012 Apr 23. PMID 22524591
- [Background] Walker EA, Shmukler C, Ullman R, Blanco E, Scollan-Koliopoulus M, Cohen HW. Results of a successful telephonic intervention to improve diabetes control in urban adults: a randomized trial. Diabetes Care. 2011 Jan;34(1):2-7. doi: 10.2337/dc10-1005. PMID 21193619
- [Derived] Levy N, Moynihan V, Nilo A, Singer K, Bernik LS, Etiebet MA, Fang Y, Cho J, Natarajan S. The Mobile Insulin Titration Intervention (MITI) for Insulin Adjustment in an Urban, Low-Income Population: Randomized Controlled Trial. J Med Internet Res. 2015 Jul 17;17(7):e180. doi: 10.2196/jmir.4716. PMID 26187303
- [Derived] Levy N, Moynihan V, Nilo A, Singer K, Bernik LS, Etiebet MA, Fang Y, Cho J, Natarajan S. The Mobile Insulin Titration Intervention (MITI) for Insulin Glargine Titration in an Urban, Low-Income Population: Randomized Controlled Trial Protocol. JMIR Res Protoc. 2015 Mar 13;4(1):e31. doi: 10.2196/resprot.4206. PMID 25794243

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Started | 33 | 28
Completed | 28 | 26
Not Completed | 5 | 2
Not completed — Phone incompatible with texting platform | 3 | 0
Not completed — Did not enroll in texting platform | 1 | 0
Not completed — Did not initiate insulin treatment | 1 | 0
Not completed — Phenotypic type 1 diabetes | 0 | 1
Not completed — Discontinued insulin - possible allergy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice | Total
Number analyzed (Participants) | 33 | 28 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.48 (11.22) | 44.61 (9.97) | 46.70 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Reach Optimal Long-acting Insulin Dose
Time Frame: 12 weeks
Population: No primary outcome data available for one participant in Current Best Practice arm who discontinued insulin early due to a mild possible allergy.
Measure: Number; unit: percentage of participants
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 33 | 27
percentage of participants | 88 | 37
Statistical Analysis 1: Comparison: Mobile Insulin Titration Intervention vs Current Best Practice; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Time to Reach Optimal Long-acting Insulin Dose
Description: The time it takes a patient to reach his/her optimal long-acting insulin dose will be measured for both study arms.
Time Frame: 12 weeks
Population: Participants who reached optimal long-acting insulin dose.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 29 | 10
weeks | 3.00 [1.29 to 4.86] | 7.07 [2.96 to 9.61]
Statistical Analysis 1: Comparison: Mobile Insulin Titration Intervention vs Current Best Practice; Test type: Superiority or Other; p = 0.007, Interval-censoring survival analysis

3. Secondary Outcome: Hemoglobin A1c
Description: Change in hemoglobin A1c
Time Frame: baseline, 12 weeks (approximately 3 months)
Population: All participants with hemoglobin A1c measurements recorded at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 28 | 14
mg/dL | -1.90 (2.64) | -1.81 (2.63)
Statistical Analysis 1: Comparison: Mobile Insulin Titration Intervention vs Current Best Practice; Test type: Superiority or Other; p = 0.99, Wilcoxon rank-sum test

4. Secondary Outcome: Baseline Treatment Satisfaction
Description: The Diabetes Treatment Satisfaction Questionnaire standard (DTSQs) will be used to measure the patient's satisfaction with diabetes treatment received prior to study participation. Scores on questionnaire range from 0 to 6: 0 = very dissatisfied, 6 = very satisfied.
Time Frame: baseline
Population: All participants who completed the treatment satisfaction questionnaire at baseline.
Measure: Mean (Standard Deviation); unit: score on satisfaction scale
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 32 | 28
score on satisfaction scale | 4.99 (1.14) | 5.20 (0.61)
Statistical Analysis 1: Comparison: Mobile Insulin Titration Intervention vs Current Best Practice; Test type: Superiority or Other; p = 0.78, Wilcoxon rank-sum test

5. Secondary Outcome: Treatment Satisfaction After Initiation of Insulin Titration
Description: The Diabetes Treatment Satisfaction Questionnaire standard (DTSQs) will be used to measure the patient's satisfaction with diabetes treatment received since initiation of long-acting insulin titration. Scores on questionnaire range from 0 to 6: 0 = very dissatisfied, 6 = very satisfied.
Time Frame: 12 weeks (approximately 3 months)
Population: All participants who completed the treatment satisfaction questionnaire at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on satisfaction scale
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 27 | 22
score on satisfaction scale | 5.74 (0.54) | 5.53 (0.52)
Statistical Analysis 1: Comparison: Mobile Insulin Titration Intervention vs Current Best Practice; Test type: Superiority or Other; p = 0.04, Wilcoxon rank-sum test

6. Secondary Outcome: Change in Treatment Satisfaction
Description: The Diabetes Treatment Satisfaction Questionnaire change (DTSQc) will be used to measure the change in the patient's satisfaction with his/her diabetes treatment since initiation of long-acting insulin titration. Scores on questionnaire range from -3 to +3: -3 = much less satisfied now, +3 = much more satisfied now.
Time Frame: 12 weeks (approximately 3 months)
Population: All participants who completed the treatment satisfaction questionnaire at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on satisfaction scale
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 27 | 22
score on satisfaction scale | 2.71 (0.71) | 2.42 (0.95)
Statistical Analysis 1: Comparison: Mobile Insulin Titration Intervention vs Current Best Practice; Test type: Superiority or Other; p = 0.13, Wilcoxon rank-sum test

7. Secondary Outcome: Incidence of Hypoglycemia
Description: The number of instances of hypoglycemia as indicated by fasting blood glucose levels or symptoms reported by patients in both study arms.
Time Frame: 12 weeks
Population: This outcome was analyzed for participants who completed the allocated intervention (and the participant who discontinued insulin early due to a mild possible allergy). Five participants reported hypoglycemia: 3 in the MITI arm and 2 in the CBP arm. All cases were mild.
Measure: Number; unit: instances of hypoglycemia
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 28 | 27
instances of hypoglycemia | 5 | 3

8. Other Pre Specified Outcome: Percentage of Text Message Responses
Description: The number of text message replies from participants compared to the total number of text messages sent to participants (asking for blood glucose values). This outcome is given as a percent.
Time Frame: 12 weeks
Population: Participants who completed the allocated intervention.
Measure: Number; unit: percentage of text messages
Units Other Than Participants: text messages sent to participants
Arm/Group | Mobile Insulin Titration Intervention
Number analyzed (Participants) | 28
Number analyzed (text messages sent to participants) | 498
percentage of text messages | 84

9. Other Pre Specified Outcome: Percentage of Successful Phone Calls
Description: The number of successful insulin titration phone calls compared to the total number of insulin titration phone calls assigned to the nurse. Successful phone calls are defined as when the nurse was able to reach the participant with one call attempt, two call attempts, or by voicemail. This outcome is given as a percent.
Time Frame: 12 weeks
Population: Participants who completed the allocated intervention.
Measure: Number; unit: percentage of phone calls
Units Other Than Participants: titration phone calls assigned to nurse
Arm/Group | Mobile Insulin Titration Intervention
Number analyzed (Participants) | 28
Number analyzed (titration phone calls assigned to nurse) | 99
percentage of phone calls | 91

10. Other Pre Specified Outcome: Patient Healthcare Utilization
Description: The number of medication refill, emergency department, and walk-in clinic visits at Bellevue Hospital (non-insulin titration visits).
Time Frame: 12 weeks
Population: All participants.
Measure: Number; unit: hospital visits
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 33 | 28
hospital visits | 6 | 11

11. Other Pre Specified Outcome: Costs - Provider Time Spent on Insulin Titration Visits
Description: Provider time spent on insulin titration visits by phone compared to insulin titration visits in the clinic.
Time Frame: 12 weeks
Population: Insulin titration visits with a duration recorded.
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: type of insulin titration visit
Groups:
- Insulin Titration Visits by Phone: Insulin titration visits that occurred over the phone in both study arms (MITI and CBP arms).
- Insulin Titration Visits in the Clinic: Insulin titration visits that occurred in the clinic in both study arms (MITI and CBP arms).
Arm/Group | Insulin Titration Visits by Phone | Insulin Titration Visits in the Clinic
Number analyzed (Participants) | 28 | 42
Number analyzed (type of insulin titration visit) | 97 | 76
minutes | 6 [3 to 10] | 30 [20 to 45]
Statistical Analysis 1: Comparison: Insulin Titration Visits by Phone vs Insulin Titration Visits in the Clinic; Test type: Superiority or Other; p = 0.008, Generalized estimating equation modeling

12. Other Pre Specified Outcome: Costs - Titration Visit Information
Description: The number of insulin titration visits (whether by phone or in the clinic).
Time Frame: 12 weeks
Population: Participants who completed the allocated intervention (and the participant who discontinued insulin early).
Measure: Median (Inter-Quartile Range); unit: insulin titration visits
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Number analyzed (Participants) | 28 | 27
insulin titration visits | 3.5 [2 to 5] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Mobile Insulin Titration Intervention vs Current Best Practice; Test type: Superiority or Other; p = 0.003, Wilcoxon rank-sum test

13. Other Pre Specified Outcome: Costs - Patient Travel Time
Description: The time it took patients to travel to Bellevue Hospital, reported by patients in both study arms at baseline and at any subsequent clinic visits.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- All Participants: Participants in both study arms (MITI and CBP).
Arm/Group | All Participants
Number analyzed (Participants) | 61
minutes | 45 [30 to 60]

14. Other Pre Specified Outcome: Costs - Co-pays
Description: At baseline, participants in both study arms (MITI and CBP) reported whether they had to pay co-pays for clinic visits at Bellevue Hospital.
Time Frame: baseline
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 61
participants | 37

15. Other Pre Specified Outcome: Qualitative Patient Satisfaction Interview
Description: The study staff will interview MITI arm patients, using free-response questions, to assess their satisfaction with the intervention. The interviews will take place in person or over the phone at the patient's convenience, after the patient has reached his/her optimal insulin dose. If the patient does not reach optimal insulin dose, the interview will take place at approximately 12 weeks.
Time Frame: After patient reaches optimal insulin dose or at 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: We were able to assess serious adverse events for participants who completed the allocated intervention (and the participant who discontinued insulin early due to a mild possible allergy). No serious adverse events were found.
Arm/Group | Mobile Insulin Titration Intervention | Current Best Practice
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 3/28 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobile Insulin Titration Intervention (N=28) | Current Best Practice (N=27)
mild hypoglycemia (General disorders) | 3 | 2
mild possible allergy to insulin (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes